CLINICAL TRIAL: NCT03705117
Title: An Open-label Exploratory Study in Patient Volunteers With Ulcerative Colitis (UC), to Investigate Lamina Propria Presence and Evidence of Biological Effect of the Oral Domain Antibody V565
Brief Title: Open-label V565 Target Engagement Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VHsquared Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: V56503
Record Dates: First submitted 2018-10-09; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V565 (Experimental): V565 orally three times daily for up to 7 days
  Interventions: Biological: V565

INTERVENTIONS:
Biological: V565 — Capsules for oral administration

SUMMARY:
The purpose of the study is to confirm that V565 enters inflamed tissue, binds to TNF and reduces inflammation after oral dosing to patients with IBD.

DETAILED DESCRIPTION:
Single-site, open-label study in up to 6 patients treated for up to 7 days with sigmoidoscopy and biopsies before and after treatment period to determine biological activity.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of UC for 12 months or more
* Distal disease, accessible by flexible sigmoidoscopy
* Mild to moderate UC as defined as Mayo score between 3 - 10 with Mayo endoscopic sub score ≥1

Exclusion Criteria:

* A known hypersensitivity to any of the inactive ingredients of the study treatment
* A diagnosis of any IBD except UC
* Isolated proctitis
* Stool culture positive for C. difficile or other enteric infection
* Untreated tuberculosis (TB); positive QuantiFERON-TB Gold Test result (performed by Central Laboratory)
* Evidence of previous or present hepatitis B or C infection
* Known severe viral infection within six weeks prior to Visit 1
* Current use of topical mesalazine or anti-infectives for serious infection (or within 1 week)
* Anti-TNFα therapy other than the study drug
* Parenteral or enteral nutrition therapy
* Current use of any biologic agent
* Primary failure or secondary loss of response (LOR) to use of a TNFα inhibitor
* Contraindication to TNFα inhibitor
* Clinically significant abnormal laboratory test result at screening
* Taken an investigational drug within 3 months or 5 half-lives (whichever is longer) prior to the first dose in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Reduction of phosphorylation in mucosal biopsies | After 7 days oral treatment
Presence of drug in mucosal biopsies | After 7 days oral treatment

CONTACTS AND LOCATIONS:
Overall Officials: Suhail Nurbhai, MBChB, Study Director — VHsquared Ltd.
Locations (1):
- The Royal London Hospital, London, United Kingdom